CLINICAL TRIAL: NCT07347184
Title: The Effect of Task-Oriented Aquatherapy Program (TOAP) on Occupational Performance and Participation in Children With Cerebral Palsy
Brief Title: The Effect of TOAP in Children With CP
Acronym: TOAP-CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aybike Baykan, Principal Investigator / Graduate Researcher, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AYBIKE-TOAP-CP-CROSSOVER-23
Record Dates: First submitted 2025-12-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP)
Keywords: aquatic therapy; occupational therapy; motivation; pool therapy; water exercise therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Two groups receive different interventions for 16 weeks, then switch interventions for another 16 weeks; each child serves as their own control.
Masking Description: Outcome evaluators (COPM, PODCI, PMOT) were blinded to group assignments to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Receives tailored occupation-based task-oriented aquatherapy program
  Interventions: Behavioral: Task-Oriented Aquatherapy Program
- Control Group (Active Comparator): Receives conventional rehabilitation exercise program
  Interventions: Other: Conventional Rehabilitation Exercise

INTERVENTIONS:
Behavioral: Task-Oriented Aquatherapy Program — A 16-week program where each child engages in activities tailored to their five most important occupations, identified via COPM. Sessions are 40 minutes, twice weekly, focused on improving occupational performance, participation, and motivation. The program is structured, individualized, and designed to enhance engagement and functional outcomes in children with CP.
  Other Names: Study Group Intervention
  Arms: Study Group
Other: Conventional Rehabilitation Exercise — Participants received standard rehabilitation exercises including activities to improve gross and fine motor skills, balance, coordination, muscle strength, joint range of motion, and cardiovascular capacity.
  Other Names: Control Group Intervention
  Arms: Control Group

SUMMARY:
This study investigates the effects of a task-oriented aquatherapy program (TOAP) on occupational performance, participation, and motivation in children with cerebral palsy. The program was designed based on each child's individually prioritized occupations identified through the Canadian Occupational Performance Measure (COPM).

Twelve children participated in a crossover design. Each child received both the TOAP intervention and conventional rehabilitation exercises in two separate 16-week periods. Interventions were delivered twice per week for 40 minutes per session. Outcomes included occupational performance (COPM), participation (PODCI), and motivation (PMOT). The study aims to provide evidence on whether personalized, meaningful, task-oriented aquatic exercises can improve functional performance and participation in children with cerebral palsy, and to offer structured TOAP protocols for clinicians.

DETAILED DESCRIPTION:
This study employed an interventional crossover desing to evaluate the effects of a task-oriented aquatherapy program (TOAP) on occupational performance, participate and motivation in children with cerebral palsy. The intervention was grounded in occupational therapy principles and structured according to the Person-Environment-Occupation (PEO) model with an emphasis on meaningful, child-selected occupations performed in an aquatic environment.

Individualized intervention goals were determined prior to the intervention using occupations prioritized by each participant through the Canadian Occupational Performance Measure (COPM). Based on these prioritized occupations, a structured TOAP was developed for each child. The program incorporated task-oriented aquatic activities designed to support functional movement, postural control, balance and engagement while emphasizing active participation and motivation during therapy sessions.

The study consisted of two consecutive 16-week intervention periods. During the first period, one group received the TOAP intervention while the comparison group received conventional rehabilitation exercises commonly used in pediatric neurorehabilitation. Following completion of the first period, the groups crossed over and received the alternate intervention in the second period. This crossover, structure allowed each participant to serve as their own control, thereby reducing inter-individual variability.

All intervention sessions were conducted twice weekly, with each sessions lasting 40 minutes. Interventions were delivered by trained clinicians in an aquatic therapy setting. Outcome assessments were conducted at baseline and at the end of the each intervention period to evaluate changes associated with each treatment condition.

The study protocol was desinged to examine whether a personalized, task-oriented aquatic intervention grounded in meaningful occupations could enhance occupational performance, participation and motivation in children with cerebral palsy and to inform the development of structured aquatic intervention approaches applicable to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Children with CP classified as GMFCS levels 1-3 and MACS levels 1-3.
* Children and caregivers who voluntarily agreed to participate

Exclusion Criteria:

* Severe intellectual disability
* MAS levels 3-4
* Surgery or botulinum toxin injection within the past 6 months
* Significant hearing or vision impairment interfering with assessment
* Medical conditions preventing exercise (e.g., cardiovascular failure)
* Conditions preventing aquatic exercise (e.g., infection, open wound, incontinence)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Occupational Performance | Baseline, up to 16 weeks (end of the first period), up to 32 weeks (end of the second period).
  Canadian Occupational Performance Measure (COPM), a client-centered outcome measure that assessing performance (COPM-Performance) in the child's top five occupations.
  Minimum value:1 Maximum value: 10 Higher score indicates greater performance.
Occupational Satisfaction with Performance | baseline, up to 16 weeks (end of the first period), up to 32 weeks (end of the second period).
  Canadian Occupational Performance Measure (COPM), a client-centered outcome measure that assessing occupational satisfaction with performance (COPM-Satisfaction) in the child's top five occupations.
  Minimum value:1 Maximum value: 10 Higher score indicates greater performance.
Participation | Baseline, up to 16 weeks (end of the first period), up to 32 weeks (end of the second period).
  Pediatric Outcomes Data Collection Instrument (PODCI) consists of six subscales. A Global Functioning Score (PODCI-GF) is calculated by summarizing the results of all six subscales. In the present study, participation and overall functional status were evaluated primarily using the PODCI-GF, as it provides a comprehensive representation of the child's overall functional participate.
  Minimum Value:0 Maximum Value:100 Higher score indicates better overall functioning

SECONDARY OUTCOMES:
Motivation | Baseline, up to 16 weeks (end of the first period), up to 32 weeks (end of the second period).
  Pediatric Motivation Scale (PMOT) consists of 19 items grouped into six subscales assessing different dimensions of motivation. A Total Motivation Score (PMOT-T) is obtained by summing the scores of all six subscales. In the present study, motivation to participate in rehabilitation programs was evaluated primarly using the PMOT-T, as it provides a comprehensive representation of the child's overall motivation toward rehabilitation.
  Minimum value:19 Maximum value: 114 Higher score indicates greater motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Sedef Şahin, Assoc. Prof., Study Director — Hacettepe University; Aybike Baykan, PT, MSc, Principal Investigator — Etimesgut Belediyesi Engelsiz Yaşam Özel Eğitim ve Rehabilitasyon Merkezi
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for each participant, including:
  COPM scores (performance and satisfaction) PODCI scores (participation) PMOT scores (motivation) Demographic information (age, sex, GMFCS and MACS levels)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available beginning 6 months after publication of the study results and will remain accessible for 5 years thereafter.
Access Criteria: Data will be accessible to qualified researchers who submit a methodologically sound proposal. Requests must be reviewed and approved by the principal investigator. Data will be shared via secure transfer under a data use agreement ensuring confidentiality and ethical use.
URL: https://www.hacettepe.edu.tr/research/datasharing

REFERENCES:
- [Result] Baykan A., Serebral Palsi Tanılı Çocuklarda Görev Odaklı Su İçi Egzersizin Okupasyonel Performans ve Katılım Üzerine Etkisi, Hacettepe Üniversitesi Sağlık Bilimleri Enstitüsü Ergoterapi Programı Yüksek Lisans Tezi, Ankara, 2023.
- See also: Hacettepe University Occupational Therapy Department Thesis Collection — https://openaccess.hacettepe.edu.tr/items/d3aac588-7d58-4c0b-bbc2-621829e4942c